CLINICAL TRIAL: NCT03599271
Title: The ASCEND Study: A Clinical Evaluation of the UP Drug-Coated Device in Patients With Chronic Rhinosinusitis
Brief Title: A Clinical Evaluation of the Intersect ENT Sinus Device (ASCEND)
Status: Completed | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: P500-0118
Record Dates: First submitted 2018-06-25; First posted 2018-07-26 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: A PK non-randomized cohort in 5 participants, followed by a randomized, intra-patient controlled double-blind cohort in 70 participants
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomized cohort is double-blinded, which both participants and outcome assessor being masked to treatment assignment
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (3):
- Drug-Coated Device (Experimental): Randomized cohort: Drug-Coated Device to dilate randomized frontal sinus ostium.
  Interventions: Device: Drug-Coated Device
- Control Sinus Dilation Device (Active Comparator): Randomized cohort: Control Device to dilate randomized contralateral frontal sinus ostium.
  Interventions: Device: Control Device
- PK cohort- Drug-Coated Device (Experimental): PK cohort: One Drug-Coated Device to dilate both frontal sinus ostia.
  Interventions: Device: Drug-Coated Device

INTERVENTIONS:
Device: Drug-Coated Device — 3000 mcg mometasone furoate-coated sinus dilation device
  Arms: Drug-Coated Device; PK cohort- Drug-Coated Device
Device: Control Device — Sinus dilation device without drug
  Arms: Control Sinus Dilation Device

SUMMARY:
The objective of the ASCEND Study is to assess the safety, performance, and efficacy of the Intersect ENT UP Drug-Coated Device when used in chronic rhinosinusitis (CRS) patients undergoing balloon dilation of frontal sinus ostia (FSO)

DETAILED DESCRIPTION:
This is a prospective, multicenter study enrolling two consecutive cohorts:

PK cohort (N=5): A non-randomized cohort to assess the systemic safety and performance of the UP Drug-Coated Device for in-office bilateral dilation of the FSO (2 inflations in each FSO for a total of 4 inflations per device). Subsequently, the UP Drug-Coated Device may be used to dilate any sphenoid or maxillary sinuses.

Randomized cohort (N=70): A randomized, intra-patient controlled, double-blind cohort of 70 subjects to assess the safety and efficacy of the UP Drug-Coated Device used for in-office dilation of the FSO. The FSO randomized to the treatment (Treatment) will undergo dilation using the UP Drug-Coated Device (2 inflations per device) while the contralateral FSO (Control) will be dilated with a UP Control Device (2 inflations per device).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CRS per the 2016, "International Consensus Statement on Allergy and Rhinology" definition.
2. Bilateral disease in the frontal sinuses (Lund-Mackay score ≥ 1 on each side) on CT scan within 30 days prior to enrollment in the PK cohort and prior to randomization in the randomized cohort.
3. Patient has bilateral obstruction of the frontal recess/FSO due to scarring and/or polypoid edema confirmed on endoscopy (patency grade of 0 or 1 for each FSO).
4. Balloon dilation of the FSO judged to be feasible and medically appropriate.
5. Patient has had prior ESS (> 30 days with a healed mucosa) including bilateral ethmoidectomy (anterior or total) and uncinectomy for better visualization of the FSO.
6. Balloon dilation of the FSO with a 6 mm balloon is judged to be feasible (use light-assisted or image-guided instrument such as a frontal sinus seeker tip to confirm access of each FSO) and medically appropriate.

Exclusion Criteria:

1. Expanded amount of ethmoid polyposis (grade > 2 PK cohort, grade ≥ 2 randomized cohort).
2. Complications from prior ESS or balloon dilation procedure (e.g., cerebrospinal fluid leak or injury to the skull base).
3. History of aspirin exacerbated respiratory disease (AERD).
4. Current smokers.
5. History of allergy or intolerance to mometasone furoate.
6. Oral-steroid dependent condition.
7. Evidence of acute rhinosinusitis, invasive fungal sinusitis or another disease or condition expected to compromise survival or ability to complete assessments during the 30-day follow-up period in the PK cohort and druing the 60-day follow-up period in the randomized cohort.
8. Use of parenteral and injected steroids (e.g., Kenalog) 30 days prior to the baseline procedure.
9. Use of oral steroids, budesonide or other sinus steroid irrigations/rinses or drops, nebulized steroids administered nasally 14 days prior to screening in the PK cohort and prior to baseline in the randomized cohort.
10. Glaucoma or posterior subcapsular cataract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centers for Advanced ENT Care, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: frontal sinuses
Groups:
- Randomized Cohort: Randomized cohort (n=70) used a randomized intra-patient design in which the Drug-Coated Device was used to dilate randomized frontal sinus ostium and Control Device was used to dilate contralateral frontal sinus ostium.
  Drug-Coated Device: 3000 mcg mometasone furoate-coated sinus dilation device. Control Device: Sinus dilation device without drug.
- PK Cohort-Safety: PK cohort (n=5) used a non-randomized design in which one Drug-Coated Device was used to dilate both frontal sinus ostia.
  Drug-Coated Device: 3000 mcg mometasone furoate-coated sinus dilation device.
Period: Overall Study
Arm/Group | Randomized Cohort | PK Cohort-Safety
Started | 70; 140 frontal sinuses | 5; 10 frontal sinuses
Drug-Coated Device | 70; 70 frontal sinuses | 5; 10 frontal sinuses
Control Device | 70; 70 frontal sinuses | 0; 0 frontal sinuses
Completed | 70; 140 frontal sinuses | 5; 10 frontal sinuses
Not Completed | 0; 0 frontal sinuses | 0; 0 frontal sinuses

BASELINE CHARACTERISTICS:
Groups:
- Randomized Cohort: Randomized cohort (n=70) used a randomized intra-patient desgin which received Drug-Coated Device to dilate randomized frontal sinus ostium and control device in the randomized contralateral frontal sinus ostium.
  Drug-Coated Device: 3000 mcg mometasone furoate-coated sinus dilation device. Control Device: Sinus dilation device without drug.
- PK Cohort- Safety: PK cohort (n=5) used a non-randomized design in which one Drug-Coated Device was used to dilate both frontal sinus ostia.
  Drug-Coated Device: 3000 mcg mometasone furoate-coated sinus dilation device.
- Total: Total of all reporting groups
Arm/Group | Randomized Cohort | PK Cohort- Safety | Total
Number analyzed (Participants) | 70 | 5 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (11.37) | 61.2 (10.94) | 54.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 1 | 27
  Male | 44 | 4 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 66 | 5 | 71
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 64 | 4 | 68
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
History of Asthma [Count of Participants; unit: Participants]
  Yes | 33 | 1 | 34
  No | 37 | 4 | 41
History of Allergic Rhinitis [Count of Participants; unit: Participants]
  Yes | 61 | 4 | 65
  No | 9 | 1 | 10
History of Aspirin Intolerance or Allergy [Count of Participants; unit: Participants]
  Yes | 2 | 1 | 3
  No | 68 | 4 | 72
History of Repeated Courses of Corticosteroids [Count of Participants; unit: Participants]
  Yes | 35 | 2 | 37
  No | 35 | 3 | 38
CT Lund Mackay Score - Total [Mean (Standard Deviation); unit: Units on a scale] — The CT Lund-Mackay score is used to assess chronic rhinosinusitis. Each sinus (frontal, anterior ethmoidal cells, posterior ethmoidal cells, maxillary sinus, and sphenoid sinus) is scored from 0 (no abnormality), 1 (partial opacification) to 2 (complete opacification). The osteomeatal complex is scored from 0 (not obstructed) to 2 (obstructed). Each side is graded separately. A combined score from 0 to 24 is possible.
  Units on a scale | 8.6 (2.94) | 11.0 (2.92) | 9.8 (2.9)
Number of Prior Endoscopic Sinus Surgery [Count of Participants; unit: Participants]
  1 | 32 | 1 | 33
  2 | 20 | 2 | 22
  3 | 10 | 0 | 10
  4 or more | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Randomized Cohort: Difference in Patency Grade of FSO
Description: Difference in the patency grade of the FSO between treatment sides at Day 30, as determined by an independent, blinded sinus surgeon based on the centralized video-endoscopy review. Patency of the FSO assessed endoscopically by probing with a 3-mm olive-shaped frontal sinus suction tip ("suction tip") and graded on a 5-point scale as follows - 0: Occluded (no opening visible); 1: Significantly stenosed (not occluded, but unable to pass the 3-mm suction tip); 2: Moderately stenosed (able to easily pass the 3-mm suction tip with no additional space around it); 3: Minimally stenosed (able to easily pass the 3-mm suction tip with additional 1-2 mm space around it); 4: Completely patent (able to easily pass the 3-mm suction tip with additional >2 mm space around it)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Randomized Cohort - Treatment Arm: Randomized cohort (n=70 patients) which received the Drug-Coated Device to dilate randomized frontal sinus ostium.
  Drug-Coated Device: 3000 mcg mometasone furoate-coated sinus dilation device
- Randomized Cohort - Control Arm: Randomized cohort (n=70) which received Control Device to dilate randomized contralateral frontal sinus ostium.
  Control Device: Sinus dilation device without drug
Arm/Group | Randomized Cohort - Treatment Arm | Randomized Cohort - Control Arm
Number analyzed (Participants) | 70 | 70
score on a scale | 1.6 (1.00) | 1.5 (1.07)

2. Primary Outcome: The Number of Participants in the PK Cohort With Successful Dilation of Attempted FSO at Baseline
Description: Successful dilation of attempted FSO using the Drug-Coated Device with no unanticipated serious adverse device effects. A successful dilation of the FSO is defined as insertion of the UP Drug-Coated Device into the targeted FSO followed by 2 consecutive, complete inflations of the balloon.
Time Frame: Baseline
Population: 'Analysis per patient.
Measure: Count of Units; unit: frontal sinus ostia
Units Other Than Participants: frontal sinus ostia
Arm/Group | PK Cohort-Safety
Number analyzed (Participants) | 5
Number analyzed (frontal sinus ostia) | 10
frontal sinus ostia | 10

3. Secondary Outcome: Randomized Cohort: Estimated Frontal Sinus Ostia (FSO) Diameter
Description: The smallest and largest diameters of the FSO determined by an independent, blinded sinus surgeon based on the centralized video-endoscopy review. FSO diameter estimated endoscopically by probing with a 3-mm olive-shaped frontal sinus suction tip and reported in mm.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Cohort - Treatment Arm | Randomized Cohort - Control Arm
Number analyzed (Participants) | 70 | 70
mm
  Largest Diameter | 2.8 (1.86) | 2.6 (1.61)
  Smallest Diameter | 2.2 (1.44) | 2.1 (1.31)

4. Secondary Outcome: PK Cohort: Estimated Largest Frontal Sinus Ostia (FSO) Diameter
Description: The smallest and largest diameters of the FSO are estimated endoscopically by probing with a 3-mm olive-shaped frontal sinus suction tip and reported in mm.
Time Frame: Baseline to 30 days
Population: Analysis per patient.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: frontal sinus ostia
Arm/Group | PK Cohort-Safety
Number analyzed (Participants) | 5
Number analyzed (frontal sinus ostia) | 10
mm
  Baseline pre-dilation | 1.2 (0.92)
  Baseline post-dilation | 3.3 (2.31)
  Day 7 | 4.1 (2.02)
  Day 14 | 3.3 (2.00)
  Day 21 | 2.4 (2.22)
  Day 30 | 2.6 (2.12)

5. Secondary Outcome: PK Cohort: Estimated Smallest Frontal Sinus Ostia (FSO) Diameter
Description: as for outcome 4
Time Frame: Baseline to 30 days
Population: Analysis per patient.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: frontal sinus ostia
Arm/Group | PK Cohort-Safety
Number analyzed (Participants) | 5
Number analyzed (frontal sinus ostia) | 10
mm
  Baseline pre-dilation | 1.1 (0.88)
  Baseline post-dilation | 2.9 (1.85)
  Day 7 | 3.2 (1.75)
  Day 14 | 3.1 (1.91)
  Day 21 | 2.1 (1.97)
  Day 30 | 2.2 (1.81)

6. Secondary Outcome: PK Cohort: Total Sino-Nasal Outcomes Test Score (SNOT-22)
Description: SNOT-22 is a validated, disease-specific, symptom-scoring instrument consisting of 22 questions, each scored by patient on a 6-point scale as follows: 0: No problem; 1: Very mild problem; 2: Mild or slight problem; 3: Moderate problem; 4: Severe problem; 5: Problem as bad as it can be.
  Sum of all 22 questions constitutes the total SNOT-22 score with a maximum total score equal to 110.
Time Frame: Baseline, Day 14 and Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PK Cohort-Safety
Number analyzed (Participants) | 5
units on a scale
  Baseline | 45.0 (10.02)
  Day 14 | 21.2 (13.9)
  Day 30 | 27.6 (9.13)

ADVERSE EVENTS:
Time Frame: 3 months
Description: In the Randomized cohort each patient received the Drug-Coated Device (Treatment Arm) and Control Device (Control Arm) and thus the adverse events were collected per patient and not per intervention.
  In the PK cohort each patient received the Drug-Coated Device only and the adverse events were collected per patient.
Groups:
- All Participants From Randomized Cohort: Randomized cohort (n=70) used a randomized intra-patient design in which the Drug-Coated Device was used to dilate randomized frontal sinus ostium and Control Device was used to dilate contralateral frontal sinus ostium.
  Each patient received the Drug-Coated Device (Treatment Arm) and Control Device (Control Arm) and thus the adverse events are reported per patient in the Randomized Cohort. The adverse events were not collected per intervention.
  Drug-Coated Device: 3000 mcg mometasone furoate-coated sinus dilation device. Control Device: Sinus dilation device without drug.
Arm/Group | All Participants From Randomized Cohort | PK Cohort-Safety
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/70 | 0/5
Other Adverse Events (participants affected / at risk) | 11/70 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants From Randomized Cohort (N=70) | PK Cohort-Safety (N=5)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants From Randomized Cohort (N=70) | PK Cohort-Safety (N=5)
Acute Sinusitis (Infections and infestations) | 11 (13) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03599271/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT03599271/SAP_001.pdf